CLINICAL TRIAL: NCT01568424
Title: CentriMag RVAS U.S. Post-approval Study Protocol
Acronym: CMagRVAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Thoratec Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TC10152008
Record Dates: First submitted 2012-03-28; First posted 2012-04-02 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Right Ventricular Failure
Keywords: Heart Failure; Right Ventricular Failure; Levitronix; Thoratec Corporation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Group (Other): Patients with acute right ventricular failure from any cause requiring use of the CentriMag RVAS to sustain life.
  Interventions: Device: CentriMag RVAS placement

INTERVENTIONS:
Device: CentriMag RVAS placement — Patients will be treated with a CentriMag RVAS

SUMMARY:
The study objective is to gather post-market clinical data on the use of the CentriMag RVAS when used for temporary mechanical circulatory support of the right ventricle in patients with acute right ventricular failure from any cause

DETAILED DESCRIPTION:
Objectives of this study are to evaluate:

1. Duration of right ventricular support
2. Incidence of adverse effects
3. Evaluation of end-organ function
4. Evaluation of hemodynamics
5. Survival at 30 days post RVAD removal

The primary endpoints include:

1. In patients who recover and do not go on to transplantation or a long-term device:

   a. Survival to 30 days post-support or to hospital discharge (whichever is longer)
2. In patients who do not recover and are bridged to transplant or a long-term system:

   1. Survival to induction of anesthesia for implantation of a long-term mechanical support device or heart transplant

Secondary endpoints include:

1. On Pump Hemodynamics

   1. A clearly observable trend toward reduction of mean right atrial pressure / central venous pressure is demonstrated while the patient is on support compared to baseline.
   2. A clearly observable trend toward an increase in mean arterial pressure is demonstrated while the patient is on support compared to baseline
   3. A clearly observable trend toward an increase in mean cardiac index is demonstrated while the patient is on support compared to baseline
2. Post Pump Hemodynamics (must meet at least two of the following criteria)

   1. Based on plotting of the data, success will be achieved if a clearly observable trend toward reduction of mean right atrial pressure/central venous pressure is demonstrated after device removal compared to baseline
   2. Based on plotting of the data, success will be achieved if a clearly observable trend toward increase in mean arterial pressure is demonstrated after device removal compared to baseline
   3. Based on plotting of the data, success will be achieved if a clearly observable trend toward increase in mean cardiac index is demonstrated after device removal compared to baseline
3. A clearly observable trend toward a reduction in creatinine and/or BUN while on support and after device removal compared to baseline
4. A clearly observable trend toward a reduction in total bilirubin while on support and after device removal compared to baseline
5. An acceptable incidence of adverse effects observed

Patient Population

This study includes data from 25 consecutive patients with acute right ventricular failure from any cause requiring use of the CentriMag RVAS to sustain life.

ELIGIBILITY:
Inclusion Criteria:

* Right ventricular failure from any cause

Exclusion Criteria:

* Primary coagulopathy or platelet disorders
* Allergy or sensitivity to heparin and all alternative anticoagulants

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-09; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Chatterjee, Study Director — Abbott Medical Devices
Locations (10):
- United States (10):
  - Mayo Clinic Hospital Arizona, Phoenix, Arizona
  - University of Kentucky, Lexington, Kentucky
  - University of Minnesota, Minneapolis, Minnesota
  - New York Columbia Presbyterian Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - St. Luke's Episcopal Medical Center, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included data from 25 consecutive patients with acute right ventricular failure from any cause requiring use of the CentriMag RVAS to sustain life. All patients implanted with a CentriMag RVAS were approached for enrollment.
Period: Overall Study
Arm/Group | Treatment Group
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This study includes data from 25 consecutive patients with acute right ventricular failure from any cause requiring use of the CentriMag RVAS to sustain life.
Arm/Group | Treatment Group
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 20
Cardiac Index (CI) [Median (Full Range); unit: L/min/m^2] | 2.4 [1.6 to 3.8]
Mean Arterial Pressure (MAP) [Median (Full Range); unit: mmHg] | 72 [59 to 106]
Central Venous Pressure (CVP) [Median (Full Range); unit: mmHg] | 11 [4 to 22]
Blood Urea Nitrogen (BUN) [Median (Full Range); unit: mg/dl] | 27 [7 to 73]
Creatinine (mg/dl) [Median (Full Range); unit: mg/dl] | 1.4 [0.5 to 4.6]
Total Bilirubin (mg/dl) [Median (Full Range); unit: mg/dl] | 1.1 [0.5 to 6.6]

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: In patients who recover and do not go on to transplantation or a long-term device: Survival to 30 days post-support or to hospital discharge (whichever is longer).
  In patients who do not recover and are bridged to transplant or a long-term system: Survival to induction of anesthesia for implantation of a long-term device or heart transplant.
Time Frame: 30 days post device removal
Measure: Number; unit: percentage of survival at 30 days
Arm/Group | Treatment Group
Number analyzed (Participants) | 25
percentage of survival at 30 days | 80

2. Secondary Outcome: Central Venous Pressure (CVP)
Description: CVP is a measure of right heart filling pressure, or the preload to the right ventricle. During RVAD support, the CVP decreases as blood is drawn into the pump and then ejected into the pulmonary artery.
Time Frame: Baseline, Day 1, Day 2, Day 3, Week 1, Prior to Explant, 1 day after RVAD removal, 2 days after RVAD removal
Population: Patients with continuous RVAD support.
Measure: Median (Full Range); unit: mmHg
Arm/Group | Treatment Group
Number analyzed (Participants) | 23
mmHg
  Baseline: number analyzed (Participants) | 20
  Baseline | 11 [4 to 22]
  Day 1 | 11 [2 to 20]
  Day 2 | 10 [6 to 24]
  Day 3: number analyzed (Participants) | 20
  Day 3 | 12 [0 to 17]
  Week 1: number analyzed (Participants) | 13
  Week 1 | 11 [0 to 16]
  Prior to explant: number analyzed (Participants) | 15
  Prior to explant | 10 [5 to 18]
  Post pump day 1: number analyzed (Participants) | 20
  Post pump day 1 | 12 [6 to 18]
  Post pump day 2: number analyzed (Participants) | 18
  Post pump day 2 | 11 [6 to 18]

3. Secondary Outcome: Mean Arterial Pressure (MAP)
Description: MAP is the mean value for the blood pressure in the arterial circulation. During RVAD support, this value provides information regarding the adequacy of cardiac output from the left ventricle.
Time Frame: Baseline, Day 1, Day 2, Day 3, Week 1, Prior to Explant, 1 day after RVAD removal, 2 days after RVAD removal.
Population: Patients with continuous RVAD support.
Measure: Median (Full Range); unit: mmHg
Arm/Group | Treatment Group
Number analyzed (Participants) | 22
mmHg
  Baseline | 72 [59 to 106]
  Day 1 | 74 [62 to 97]
  Day 2: number analyzed (Participants) | 21
  Day 2 | 74 [55 to 104]
  Day 3: number analyzed (Participants) | 21
  Day 3 | 75 [62 to 105]
  Week 1: number analyzed (Participants) | 16
  Week 1 | 79 [54 to 90]
  Prior to explant: number analyzed (Participants) | 20
  Prior to explant | 77 [62 to 94]
  Post pump day 1: number analyzed (Participants) | 20
  Post pump day 1 | 73 [60 to 82]
  Post pump day 2: number analyzed (Participants) | 20
  Post pump day 2 | 72 [62 to 87]

4. Secondary Outcome: Cardiac Index (CI)
Description: Cardiac output (L/min) divided by the body surface area (m2)
Time Frame: Baseline, Day 1, Day 2, Day 3, Week 1, Prior to Explant, 1 day after RVAD removal, 2 days after RVAD removal.
Population: Patients with continuous RVAD support
Measure: Median (Full Range); unit: L/min/m2
Arm/Group | Treatment Group
Number analyzed (Participants) | 9
L/min/m2
  Baseline | 2.4 [1.6 to 3.8]
  Day 1 | 2.2 [1.7 to 5.6]
  Day 2: number analyzed (Participants) | 7
  Day 2 | 2.9 [1.6 to 5.6]
  Day 3: number analyzed (Participants) | 6
  Day 3 | 3.0 [1.8 to 4.5]
  Week 1: number analyzed (Participants) | 1
  Week 1 | 7.7 [7.7 to 7.7]
  Prior to explant: number analyzed (Participants) | 5
  Prior to explant | 2.7 [1.8 to 4.2]
  Post pump day 1: number analyzed (Participants) | 7
  Post pump day 1 | 2.2 [1.8 to 3.0]
  Post pump day 2: number analyzed (Participants) | 8
  Post pump day 2 | 2.3 [1.9 to 3.4]

5. Secondary Outcome: Blood Urea Nitrogen (BUN)
Description: BUN is a measure of renal function
Time Frame: Baseline, Day 1, Day 2, Day 3, Week 1, Prior to Explant, 1 day after RVAD removal, 2 days after RVAD removal, 30 days after RVAD removal
Population: Patients with continuous RVAD support
Measure: Median (Full Range); unit: mg/dl
Arm/Group | Treatment Group
Number analyzed (Participants) | 25
mg/dl
  Baseline | 27 [7 to 73]
  Day 1: number analyzed (Participants) | 23
  Day 1 | 27 [9 to 71]
  Day 2: number analyzed (Participants) | 23
  Day 2 | 26 [9 to 95]
  Day 3: number analyzed (Participants) | 22
  Day 3 | 33 [8 to 109]
  Week 1: number analyzed (Participants) | 16
  Week 1 | 28 [9 to 101]
  Prior to explant: number analyzed (Participants) | 21
  Prior to explant | 22 [10 to 67]
  Post pump day 1: number analyzed (Participants) | 20
  Post pump day 1 | 28 [12 to 72]
  Post pump day 2: number analyzed (Participants) | 19
  Post pump day 2 | 31 [14 to 79]
  30 days: number analyzed (Participants) | 19
  30 days | 24 [7 to 123]

6. Secondary Outcome: Creatinine
Description: Creatinine is a measure of renal function
Time Frame: as for outcome 5
Population: Patients with continuous RVAD support
Measure: Median (Full Range); unit: mg/dl
Arm/Group | Treatment Group
Number analyzed (Participants) | 25
mg/dl
  Baseline | 1.4 [0.5 to 4.6]
  Day 1: number analyzed (Participants) | 23
  Day 1 | 1.3 [0.6 to 3.7]
  Day 2: number analyzed (Participants) | 23
  Day 2 | 1.1 [0.6 to 4.8]
  Day 3: number analyzed (Participants) | 22
  Day 3 | 1.2 [0.5 to 5.2]
  Week 1: number analyzed (Participants) | 16
  Week 1 | 1.0 [0.6 to 4.5]
  Prior to explant: number analyzed (Participants) | 21
  Prior to explant | 1.0 [0.6 to 2.8]
  Post pump day 1: number analyzed (Participants) | 20
  Post pump day 1 | 1.2 [0.6 to 3.7]
  Post pump day 2: number analyzed (Participants) | 19
  Post pump day 2 | 1.3 [0.4 to 4.2]
  30 days: number analyzed (Participants) | 19
  30 days | 1.3 [0.6 to 5.5]

7. Secondary Outcome: Total Bilirubin
Description: Total bilirubin is a measure of hepatic function
Time Frame: as for outcome 5
Population: Patients with continuous RVAD support
Measure: Median (Full Range); unit: mg/dl
Arm/Group | Treatment Group
Number analyzed (Participants) | 24
mg/dl
  Baseline | 1.1 [0.5 to 6.6]
  Day 1: number analyzed (Participants) | 19
  Day 1 | 3.0 [0.6 to 3.7]
  Day 2: number analyzed (Participants) | 21
  Day 2 | 3.0 [0.3 to 7.1]
  Day 3: number analyzed (Participants) | 18
  Day 3 | 2.8 [0.9 to 12.3]
  Week 1: number analyzed (Participants) | 13
  Week 1 | 1.8 [0.7 to 6.4]
  Prior to explant: number analyzed (Participants) | 16
  Prior to explant | 1.3 [0.2 to 10.4]
  Post pump day 1: number analyzed (Participants) | 17
  Post pump day 1 | 2.0 [0.7 to 9.9]
  Post pump day 2: number analyzed (Participants) | 13
  Post pump day 2 | 1.3 [0.4 to 7.0]
  30 days: number analyzed (Participants) | 10
  30 days | 0.8 [0.2 to 7.2]

ADVERSE EVENTS:
Time Frame: Baseline through 6 month follow-up
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 7/25
Serious Adverse Events (participants affected / at risk) | 24/25
Other Adverse Events (participants affected / at risk) | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=25)
Infection (Infections and infestations) | 13 (23)
Bleeding (Blood and lymphatic system disorders) | 16 (40)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 16 (19)
Arrhythmias (Cardiac disorders) | 13 (14)
Hypertension (Cardiac disorders) | 5 (9)
Hepatic Dysfunction (Hepatobiliary disorders) | 0 (0)
Renal Failure (Renal and urinary disorders) | 11 (11)
Neurologic Dysfunction (Stroke) (Nervous system disorders) | 4 (4)
Thrombotic Vascular (Vascular disorders) | 1 (1)
Pericardial Fluid Collection (Cardiac disorders) | 4 (5)
Right Heart Failure (Cardiac disorders) | 6 (7)
Hemolysis (Blood and lymphatic system disorders) | 2 (2)
Device Failure (Product Issues) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Psychiatric Episode (Psychiatric disorders) | 1 (1)
Arterial non-CNS (Vascular disorders) | 1 (1)
Other (General disorders) | 7 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other